CLINICAL TRIAL: NCT03915197
Title: Risk of Allergic Asthma Occurring in the Long Term From an Episode of Acute Bronchiolitis in Infants: Clinical, Allergological and Functional Evaluation in the Long Term
Brief Title: Acute Bronchiolitis in Infants and Allergic Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-433; 2018-A02659-46 (Other: 2018-A02659-46)
Record Dates: First submitted 2019-04-01; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Acute Bronchiolitis; Asthma; Allergy
Keywords: allergic asthma; acute bronchiolitis; allergic sensitization; -risk factor
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group 1 (Experimental): cohorts of infants with acute bronchiolitis
  Interventions: Diagnostic Test: Pneumological evaluation

INTERVENTIONS:
Diagnostic Test: Pneumological evaluation — Consultation with a pneumopediatrician: collection of respiratory symptoms, respiratory treatments, evaluation of the atopic site and environmental risk factors for bronchial aggression, especially passive smoking

SUMMARY:
Predicting the risk of allergenic sensitizations and asthma development in the first year of life is difficult.

Investigator decided to follow prospectively two cohorts of infants with acute bronchiolitis, hospitalized or treated at home, from the epidemic seasons of 2011-2012 and 2015-2017 to know their respiratory evolution, especially if they developed allergen sensitization and / or asthma.

DETAILED DESCRIPTION:
Follow-up consultation 6 years after an episode of acute bronchiolitis at Clermont-Ferrand hospital with:

* Consultation with a pneumopediatrician: collection of respiratory symptoms, respiratory treatments, evaluation of the atopic site and environmental risk factors for bronchial aggression, especially passive smoking;
* Physical examination ;
* Evaluation of precariousness during the same interview with the EPICES questionnaire;
* Prick tests with positive control (histamine) and negative (physiological saline) and prick for the main pneumallergens (mites, alternaria, grasses, cat and dog) and trophallergens (egg, milk, fish, soy, wheat, peanut);
* Blood test with blood count, determination of specific IgE (5 pneumallergens and 5 trophallergens), dosage of sRAGE;
* Fonctionnal respiratory test with reversibility test

ELIGIBILITY:
Inclusion Criteria:

- Acute bronchiolitis in an infant less than one year old, included in studies KL6 (winter period 2011-2012) or CC16 (winter period 2015-2016) at clermont-ferrand hospital.

Exclusion Criteria:

* Bronchopulmonary dysplasia;
* History of prematurity <34 AS;
* Mucoviscidosis;
* known immune deficiencies;
* Primary ciliary dyskinesia suspected;
* Congenital heart disease;
* Acute renal failure.
* Refusal of parents to participate

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2019-05-02 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Risk factors for asthma 6 years after an episode of acute bronchiolitis | at 6 years
  Presence / absence of asthma 6-9 years after an episode of bronchiolitis during the first year of life
  The diagnosis of asthma is established during a consultation by a pneumopediatrician on the following criteria:
  * ≥3 documented respiratory symptoms ≥ 2 times;
  * Or an episode lasting ≥ 4 weeks;
  * With symptoms: tachypnea, wheezing, expiratory stridor, signs of chest retraction or wheezing diagnosed by a doctor.

SECONDARY OUTCOMES:
Correlation between onset of asthma and severity of bronchiolitis | at 6 years
  Severity of acute bronchiolitis, assessed by a clinical score based on control signs, spO2 and respiratory rate (Wainwright score) and the length of hospital stay
relationship between KL-6 serum markers and the occurrence of longer-term asthma | at 6 years
  Correlation between onset of asthma and concentration of KL-6 during bronchiolitis
relationship between CC16 serum markers and the occurrence of longer-term asthma | at 6 years
  Correlation between onset of asthma and concentration of CC16 during bronchiolitis.
relationship between sRAGE serum markers and the occurrence of longer-term asthma | at 6 years
  Correlation between onset of asthma and concentration of sRAGE during bronchiolitis

CONTACTS AND LOCATIONS:
Overall Officials: André LABBE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France